CLINICAL TRIAL: NCT03693937
Title: A Retrospective Registry Study to Evaluate the Long-Term Efficacy and Safety of Superficial Radiation Therapy (SRT) in Individuals With Non-Melanoma Skin Cancer (NMSC) .
Brief Title: A Retrospective Evaluation of Superficial Radiation Therapy (SRT) and Non-Melanoma Skin Cancer (NMSC)
Status: Completed | Type: Observational
Sponsor: Sensus Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: SRTS-SRT-001
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-04

CONDITIONS: Non-melanoma Skin Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Radiation: SRT-100 — The SRT-100™ is a simple painless non-invasive in-office procedure that is approved by the U.S. Food and Drug Administration (U.S. FDA) to treat keloids caused by surgery or injury by delivering a precise, calibrated dose of Superficial Radiation Therapy (SRT) that only goes skin deep.

SUMMARY:
Non-Melanoma Skin Cancer (NMSC) is the most commonly occurring type of skin cancer, and predominantly comprises (98%) Basal Cell Carcinomas (BCC) and Squamous Cell Carcinomas (SCC). About 3.3 million people in the United States (U.S.) are diagnosed with NMSC annually, equating about 5.4 million BCCs and SCCs. Low-dose Superficial Radiation Therapy (SRT) effectively destroys BCC and SCC without any invasive cutting, bleeding or stitching. There is no need for anesthesia, no risk of infection or scarring and no need for reconstructive plastic surgery. Healing time is quick with minimal to no post-treatment downtime or lifestyle restrictions. It is therefore both a viable and highly desirable alternative to invasive, painful and higher-risk surgical procedures. This study will utilize retrospective chart analysis to evaluate the outcomes of SRT-100™ therapy on NMSC lesions over a long-term post-treatment period.

DETAILED DESCRIPTION:
Non-Melanoma Skin Cancer (NMSC) is the most commonly occurring type of skin cancer and accounts for about one-third of all cancers. NMSCs predominantly (98%) include Basal Cell Carcinomas (BCC) and Squamous Cell Carcinomas (SCC). Basal cell carcinomas (BCC) are abnormal, uncontrolled growths or lesions that arise in the skin's basal cells that line the deepest layer of the epidermis, occurring most commonly on sun-exposed areas of the face, head and neck. They are slow-growing cancers that rarely metastasize. Delayed or ineffective treatment of BCCs can lead to disfigurement of the lesion and recurrence. Squamous cell carcinomas (SCC) are uncontrolled growths of abnormal cells arising from the squamous cells in the epidermis producing keratin, also typically developing on sun-exposed and damaged body areas such as the face, ears, neck, lips, back of the hands, arms and legs. SCCs may be slow or rapidly growing with significant tenderness and pain and may become disfiguring and fatal if left untreated and allowed to grow.

About 3.3 million people in the United States (U.S.) are diagnosed with NMSC annually, equating about 5.4 million BCCs and SCCs. Diagnosis and treatment of NMSC in the U.S. increased by 77% between 1994 and 2014. The incidence of BCC is about 4 times that of SCC. An estimated 4.3 million cases of BCC are diagnosed annually in the U.S. resulting in over 3,000 deaths. Over 1 million cases of SCC are diagnosed in the U.S. annually, resulting in over 15,000 deaths. SCC has a 4% annual incidence of metastasis. About 90% of NMSC is associated with repeated and unprotected skin exposure to ultraviolet (UV) rays

Treatment options for NMSC include surgery, cryotherapy, curettage and electrodesiccation, radiation therapy including superficial radiation therapy (SRT), photodynamic therapy, various forms of brachytherapy, and chemotherapeutic agents.

Low-dose SRT effectively destroys BCC and SCC without any invasive cutting, bleeding or stitching. There is no need for anesthesia, no risk of infection or scarring and no need for reconstructive plastic surgery. Healing time is quick with minimal to no post-treatment downtime or lifestyle restrictions. It is therefore both a viable and highly desirable alternative to invasive, painful and higher-risk surgical procedures. This study will utilize retrospective chart analysis to evaluate the outcomes of SRT-100™ therapy on NMSC lesions over a long-term post-treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with SRT-100™.
* Treatment date of December 31, 2015 or earlier.
* Non-Melanoma Skin Cancer (NMSC) pathological diagnosis of confirmed squamous cell carcinoma (SCC) or basal cell carcinoma (BCC).
* Histopathological Grade: G1 (well differentiated); G2 (moderately differentiated) or Gx (not assessed).
* One lesion is treated, or more than one lesion is treated with a minimum of a 5 mm gap between the edges of the lesion margins.
* Required retrospective data is existing and sufficient.

Exclusion Criteria:

* Lesions of etiology other than non-melanoma skin cancer (NMSC)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population comprises patients who were treated with the SRT-100™ for one or more non-melanoma skin cancers (NMSCs) and have follow-up data.
Sampling Method: Non-Probability Sample
Enrollment: 776 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-03-16 (Actual); Study Completion 2019-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Roth, M.D., Principal Investigator
Locations (1):
- Dermatology and Dermatological Surgery, Boynton Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-Melanoma Skin Cancers (NMSCs): Non-Melanoma Skin Cancers (NMSCs) treated with SRT-100 therapy.
Period: Overall Study
Arm/Group | Non-Melanoma Skin Cancers (NMSCs)
Started | 776
Completed | 776
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Non-Melanoma Skin Cancers (NMSCs)
Number analyzed (Participants) | 516
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.94 (8.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 223
  Male | 293
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Participant Race: Hispanic or Latino | 0
  Participant Race: Not Hispanic or Latino | 516
  Participant Race: Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 516

OUTCOME MEASURES:

1. Primary Outcome: Cure Rate
Description: NMSC cure rate will be calculated as the percentage of lesions that attained complete cure following SRT-100 treatment completion.
Time Frame: 5 years
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Non-Melanoma Skin Cancers (NMSCs)
Number analyzed (Participants) | 776
Number analyzed (lesions) | 760
lesions | 751

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Non-Melanoma Skin Cancers (NMSCs)
All-Cause Mortality (participants affected / at risk) | 0/776
Serious Adverse Events (participants affected / at risk) | 0/776
Other Adverse Events (participants affected / at risk) | 6/776
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Melanoma Skin Cancers (NMSCs) (N=776)
Radiation Dermatitis (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/37/NCT03693937/Prot_SAP_000.pdf